CLINICAL TRIAL: NCT05906069
Title: ITreatOCD: Predicting the Efficacy of Internet-based Cognitive Behavioral Therapy from Changes in the Neurobiological Correlates of Emotion Regulation in Obsessive-compulsive Disorder
Brief Title: ITreatOCD: Predicting the Efficacy of Internet-based Cognitive Behavioral Therapy in Obsessive-compulsive Disorder
Acronym: iTREATOCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pedro Morgado (Other)
Collaborators: Hospital de Braga (Other); ICVS - Life and Health Sciences Research Institute (Unknown); Clinical Academic Center (2CA) (Unknown); Associação Centro de Medicina P5 (ACMP5) (Unknown)
Responsible Party: Sponsor-Investigator, Pedro Morgado, Assistant Professor, M.D., Ph.D., University of Minho
Organization: University of Minho (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iTREATOCD_ICVS2022
Record Dates: First submitted 2023-05-16; First posted 2023-06-15 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: obsessive-compulsive disorder; ocd; neuroimaging; emotion regulation; internet-based cognitive behavioral therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Compulsive Personality Disorder; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: OCD patients will be randomly allocated into two groups - iCBT group (experimental group) and wait list group (comparator control group). The experimental group will receive a 14-week iCBT intervention program and the wait list group will receive the same intervention but at a later time.
Who Masked: Outcomes Assessor
Masking Description: The psychologist performing the assessment of the main psychometric outcomes will be blind to the group allocation of each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iCBT intervention (Experimental): Participants will enroll in an internet-based cognitive behavioral program during 14 weeks. The program comprises 10 modules and three videoconferencing psychotherapy sessions.
  Interventions: Behavioral: ICBT
- Wait list (No Intervention): Participants will be enrolled in the iCBT program after 14 weeks

INTERVENTIONS:
Behavioral: ICBT — The intervention will consist in a structured internet-based intervention with 10 modules that will combine cognitive-behavioral techniques to improve obsessive-compulsive symptoms as well as the emotion regulation ability.
  Arms: iCBT intervention

SUMMARY:
In the current study, the investigators will characterize obsessive-compulsive disorder (OCD) patients and healthy controls with a comprehensive clinical and neuroimaging assessment, focusing on the basic psychological processes related and on the neurobiological underpinnings of emotion regulation (ER). After a baseline assessment, the investigators will implement an internet-based cognitive behavioral therapy (iCBT) protocol and assess its efficacy on the modulation of ER and OCD severity. Specifically, the investigators will (1) examine to what extent the iCBT intervention modulates ER and the associated neurobiological mechanisms and (2) identify candidate biomarkers of successful treatment response.

DETAILED DESCRIPTION:
Sixty patients and sixty controls will be recruited at Hospital de Braga, Braga, Portugal (sample size estimated based on a previous systematic review). A power analysis indicated that a sample of 24 individuals per group is adequate to detect an effect size of d=.89, with a Type I error of .05 and a statistical power of .85. A final sample of 30 individuals was defined to account for a 20% dropout rate during the intervention.

All participants will be assessed with a comprehensive psychological and clinical characterization. Following the baseline assessment, OCD patients will be randomly allocated to the intervention (iCBT intervention) or the control group (waiting list). The iCBT intervention will consist of a structured program comprising 10 modules with text and video content, as well as 3 videoconferencing psychotherapy sessions. After the intervention/waiting list, patients will be re-assessed with the clinical and psychological assessment.

In order to characterize the patterns of brain activation in OCD patients during an emotion regulation task in comparison to healthy controls and to identify potential neurobiological markers of symptoms' improvement, a multimodal neuroimaging assessment will also be performed. The task encompasses the presentation of pictures (fearful, neutral and OCD-related stimuli) under two conditions: the instruction to view the pictures naturally ('observe'); or to apply cognitive reappraisal techniques to decrease any negative affective state caused by the stimuli ('regulate'). Fear and OCD-related pictures are presented during both conditions; neutral pictures only during 'observe'. After each stimulus, the level of distress will be assessed by a self-report rating scale.

In the baseline assessment, brain activation patterns (with whole-brain and region of interest approaches) will be compared between OCD and healthy controls in both task conditions. After intervention, emotion regulation ability and the underlying neurobiological mechanisms will be compared between the 'intervention' and 'waiting list' groups.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of current OCD according to the fifth Diagnostic and Statistical Manual of Mental Disorders
* YBOCS score ≥ 16
* Psychotropic medication, if stable for at least 2 months prior to inclusion and if the dosage is maintained thoughout the study
* Have the resources to access the online intervention (internet access; computer or tablet)

Exclusion Criteria:

* MRI contraindications
* Prior medical history of neurological disorders or traumatic brain injury
* Having performed CBT treatment for OCD in the last 2 years
* Undergoing any psychological treatment
* Suicidal ideation
* Current alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | immediately before and immediately after intervention/waitlist
  Psychometric scale to assess obsessive-compulsive symptoms

SECONDARY OUTCOMES:
Obsessive-Compulsive Inventory- Revised | baseline; 4 weeks after beginning intervention/waitlist; 8 weeks after beginning; 12 weeks after beginning intervention/waitlist and immediately after intervention/waitlist
  Psychometric scale to assess obsessive-compulsive symptoms
Hamilton Anxiety Scale | immediately before and immediately after intervention/waitlist
  Psychometric scale to assess anxiety symptoms
Hamilton Depression Scale | immediately before and immediately after intervention/waitlist
  Psychometric scale to assess depression symptoms
Perceived Stress Scale | immediately before and immediately after intervention/waitlist
  Psychometric scale to assess stress symptoms
Emotion Regulation Questionnaire | immediately before and immediately after intervention/waitlist
  Psychometric scale to assess cognitive regulation and emotional suppression capabilities
Difficulties in Emotion Regulation Scale | immediately before and immediately after intervention/waitlist
  Psychometric scale to assess emotion deregulation
Positive and Negative Affect Schedule | immediately before and immediately after intervention/waitlist
  Psychometric scale to assess affect
Depression Anxiety Stress scale | baseline; every week during intervention/wait list (up to 14 weeks) and immediately after intervention/waitlist
  Psychometric scale to assess symptoms of anxiety, depression and stress
NEO Five-Factor Inventory | baseline
  Psychometric scale to assess personality traits
Treatment Acceptability/Adherence Scale | immediately after intervention
  Psychometric scale to assess treatment adherence
University of Rhode Island Change Assessment Scale | baseline
  Psychometric scale to assess motivation to change

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Morgado, M.D, Ph.D., Principal Investigator — Life and Health Sciences Research Institute (ICVS), School of Medicine, University of Minho
Locations (1):
- Life and Health Sciences Research Institute, School of Medicine, University of Minho, Braga, Gualtar, Portugal

IPD SHARING:
Plan to Share IPD: No